CLINICAL TRIAL: NCT05379374
Title: Comparison of Analgesic Effects of Ultrasound Guided Transversus Abdominis Plane Block With Bupivacaine and Bupivacaine With Morphine in Patient Undergoing Open Unilateral Inguinal Hernia Repair Under Spinal Anaesthesia
Brief Title: Effects of Morphine Added to Bupivacaine in Transversus Abdominis Plane Block for Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, Purna Kala Gurung, Principal Investigator ( Assistant Professor), B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRC/1182/017
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Inguinal Hernia
Keywords: TAP block,; Morphine,; Inguinal hernia
MeSH Terms: conditions — Hernia, Inguinal | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Intervention Model Description: After obtaining written informed consent from a total of 40 patients fulfilling inclusion criteria will be enrolled. A 40 envelopes with number indicating the sequence of the patient on the outside and the allocated group and study drug inside will be made by an anaesthesiologist. An anaesthetic technician will prepare the study drug. The participants, clinicians and the investigator who is involved in patient assessment and collecting data postoperatively will be blinded.
  The study groups received the following study medication Group B - 0.25% bupivacaine 20 ml in TAP block Group BM - 0.25% bupivacaine 20 ml with 3 mg morphine in TAP block
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Anaesthetic technician will prepare the study drug
  * Anaesthesiologist who is blind to the study drug will perform UG TAP block and collect data intra and post-operatively.
  * Patient will also be blind about the drug administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine group (Active Comparator): 0.25% bupivacaine 20 ml in TAP block
  Interventions: Combination Product: bupivacaine and morphine
- Bupivacaine morphine group (Experimental): 0.25% bupivacaine 20 ml with 3 mg morphine in TAP block
  Interventions: Combination Product: bupivacaine and morphine

INTERVENTIONS:
Combination Product: bupivacaine and morphine — Bupivacaine group will receive 0.25% bupivacaine 20 ml in TAP block. Bupivacaine morphine group will receive 0.25% bupivacaine 20 ma with 3 mg morphine in TAP block.

SUMMARY:
This study is conducted to determine whether morphine added to bupivacaine in ultrasound guided (USG) transversus abdominis plane (TAP) block has beneficial effects than bupivacaine alone in providing postoperative analgesia for inguinal hernia surgery.

DETAILED DESCRIPTION:
Total of forty adult patients of American Society of Anaesthesiologists (ASA) physical status ( PS) I - II scheduled for elective inguinal hernia surgery under spinal anaesthesia were recruited in this study after getting written informed consent. They were randomized to undergo ipsilateral USG TAP block with 20 ml of 0.25 % bupivacaine (group B) versus 20 ml of 0.25 % bupivacaine with 3 mg morphine (group BM). Patients were followed postoperatively for the 24 hours by a blinded investigator for monitoring of number of rescue analgesic consumed, duration of analgesia, numerical rating scale (NRS) at rest and on cough and any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

ASA I to III Elective surgery

Exclusion Criteria:

* Patient's refusal
* BMI > 35 kg/m2 or < 18 kg/m2
* Allergic or contraindication to drugs used in study
* Coagulopathy
* Local site infection
* Spine deformity
* Uncooperative or psychological illness
* Inability to comprehend pain scale
* Drugs not injected in target area

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-08-18 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
• Duration of postoperative analgesia • Postoperative analgesic requirement | Till 24 hour after surgery
  Time from TAP block to first request of analgesic is considered as duration of analgesia Less requirement of rescue analgesic is considered as better

SECONDARY OUTCOMES:
• NRS for pain at rest and on cough between the groups • Any side effects | Till 24 hour after surgery
  Group with higher NRS score is considered a less effective Group with increase side effects is considered as not acceptable

CONTACTS AND LOCATIONS:
Overall Officials: Purna k Gurung, MS, Principal Investigator — B.P. Koirala Institute of Health Sciences
Locations (1):
- Purna kala Gurung, Dharān, Province No. 1, Nepal

IPD SHARING:
Plan to Share IPD: No